CLINICAL TRIAL: NCT06143228
Title: The Influence of Directional Preference on Movement Coordination Deficits in Individuals With Whiplash Associated Disorders
Brief Title: Influence of Directional Preference on Movement Coordination Deficits in Individuals With Whiplash Associated Disorders
Status: Recruiting | Type: Observational
Sponsor: D'Youville College (Other)
Responsible Party: Sponsor
Other Study IDs: 081469
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Whiplash Injury of Cervical Spine; Muscle Weakness
Keywords: Whiplash Associated Disorders; Movement Coordination Deficits; McKenzie; Neck Pain
MeSH Terms: conditions — Muscle Weakness; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Whiplash Associated Disorder with Directional Preference: Movements that reduce, abolish, or centralize the patient symptoms are recognized as a directional preference. Directional preference is ultimately used to guide the treatment of neck pain related to derangement syndrome.If the patient neck impairments are related to a Derangement syndrome, the patient will be instructed to perform the movements in the identified directional preference every 2-3 hours for 10-12 repetitions or to hold the cervical spine in a sustained position for 1-2 minutes. If the response to the intervention plateaus, the exercise intensity is progressed through the application of patient self-overpressure. If warranted clinician overpressure and mobilization may be utilized as a progression beyond patient generated forces. to achieve a favorable response.
- Whiplash Associated Disorder without Direction Preference: Patients with WADs that do not demonstrate directional preference will be managed based on the published Clinical Practice Guidelines (2017) for management of WADs with related movement coordination deficits. Treatment and progression of care for this group will be determined by the treating therapist but will consist of education, multimodal care inclusive of therapeutic exercise, mobilization, aerobic exercise, flexibility, and postural education. In addition, if the patient symptoms are chronic in nature treatment may include exercise progression, education and reassurance, transcutaneous nerve electrical stimulation, and cognitive behavioral therapy are recommended.

SUMMARY:
The aim of this prospective observational study is to investigate whether the presence or absence of directional preference impacts movement coordination impairments as measured in patients with Whiplash Associated Disorders (WAD).

The primary research question this study aims to answer is:

1. Is the presence of directional preference in patients with WADs associated with more favorable improvements in the specific outcome measures as compared to those patients with WADs without the presence of directional preference.

Patients in this study will asked to complete the following measures at baseline, during care, discharge, and 3 month follow up.

1. Numeric Pain Rating Scale (NPRS)
2. Optimal Screening for Prediction and Referral and Outcome-Yellow Flag (OSPRO-YF)
3. Neck Disability Index (NDI)
4. Craniocervical Flexion Test (CCFT)
5. Neck Flexor Endurance Test
6. Cervical Range of Motion

Patients demonstrating a directional preference will be managed utilizing a Mechanical Diagnosis and Treatment approach (MDT) while those without directional preference will be managed according to published clinical practice guidelines for patients with Neck Pain and Movement Coordination Deficits (WADs).

DETAILED DESCRIPTION:
Objective The primary aim of this prospective observational study is to investigate whether the presence or absence of directional preference impacts movement coordination impairments as measured at the start of care, during care, discharge, and at 3 month follow up. It is hypothesized that the presence of directional preference in patients with WADs may be associated with more favorable improvements in the specific outcome measures as compared to the group without the presence of directional preference.

Design: Prospective Observation Cohort Design

Background: Neck pain ranks 19th in global disability-adjusted life years with an overall prevalence of 27 per 1000 population with variation based on geographic location amongst other factors. The clinical course of neck pain is variable and not always favorable. A research dearth remains in whiplash associated disorders (WAD) and movement coordination issues for the cervical spine.

Movement coordination impairments are commonly associated with whiplash associated disorders. Poorer prognosis is associated with older age, higher initial neck disability index, high initial pain intensity. Recovery slows down after the first 6-12 weeks, and some patients have with persistent pain and disability even 1 year after the whiplash associated disorder. However, the prognostic value of limited cervical mobility and altered motor control has also been questioned. The use of mechanical diagnosis and therapy (MDT) has been associated with better function, range of motion, and overall lower costs in whiplash associated disorders at both the 6 and 36 month mark but whether the results differ from natural history or other approaches is debatable.

Setting:

The settings for subject recruitment and all data collection are two outpatient physical therapy clinics located in the southeastern United States during the period of September 2023 to September 2024. Prior approval for data collection will be obtained in writing from the clinic directors of both sites.

Sample and Population:

Convenience sampling will be utilized for this study. A G-power a priori power analysis with a medium effect size determined that a sample size of 55 is required to achieve a statistical power of .80 with an alpha level of .05. A total of 65 subjects will be recruited between the two data collection sites to account for an expected 20% attrition rate on follow up.

Procedures: Subjects referred to one of two out-patient physical therapy clinics meeting inclusion criteria will be evaluated, classified using a Mechanical Diagnosis and Treatment (MDT) approach. Those patients demonstrating a directional preference will be managed using an MDT approach while those not demonstration a directional preference will be managed using published clinical practice guidelines for patients with Movement Coordination Deficits (WADs). Outcome measures will be taken at baseline, visit 5, visit 10 or discharge (whichever comes first) and 3 month follow up.

Data Analyses:

Descriptive statistics will be used to assess patient baseline and change scores on the dependent variables of interest. Inferential statistics (linear regression) will be utilized to assess for statistically significant changes over time and between groups for the variables of interest.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-70
* Symptom complaints are related to a motor vehicle collision or trauma.
* Pain presents as unilateral or bilateral head/neck, upper back, or arm pain and/or stiffness
* Patient has been previously screened by their MD and received appropriate imaging to rule out the possibility of cervical fracture.

Exclusion Criteria:

* Neck pain is determined to be of non-cervical origin
* Malignancy/infection
* Presence of progressive neurological deficits
* Cranial or cervical vascular disorder
* Substance use or withdrawal
* Acute post cervical surgery
* Psychosis/psychiatric disorder/post-traumatic stress disorder
* Vertigo with nystagmus is present

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of interest for this study will consist of subjects meeting inclusion criteria referred by their physician to one of two out-patient physical therapy clinics located in the southwestern United States.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Craniocervical Flexion Test (CCFT) | Baseline, 3 weeks, 6 weeks
  Measures the holding capacity of the deep cervical flexor muscles: longus capitis and longus coli.To measure the deficit, an inflatable pressure biofeedback device (Stabilizer, Chattanooga, Tennessee, USA) is placed behind the patient's neck while the patient is hook-lying in the supine position. The pressure sensor is inflated to a baseline pressure of 20 mmHg. The patient is then instructed to perform head nodding motions of craniocervical flexion. The patient is instructed to hold a head-nodding motion for ten seconds at a baseline of 20 mmHg. After this step, the patient's pressure is progressively increased by 2 mmHg in 10 second intervals until a maximum of 30 mmHg is achieved. If the patient failed to maintain the head-nodding position at a certain pressure, then the measurement is recorded.
Neck Flexor Endurance Test: | Baseline, 3 weeks, 6 weeks
  Used to measure the holding capacity of the deep cervical flexor muscles. The participant was instructed to tuck their chin, lift their head off the table, and hold that position until exhaustion, or onset of symptoms. The physical therapist administering the test used a stopwatch to assess duration of hold. The test was concluded if the patient demonstrated any of the following: protrusion, shaking, onset or worsening of symptoms, or touching the table with their head.18, neck pain versus no neck pain.
Cervical Range of Motion (CROM) | Baseline, 3 weeks, 6 weeks
  A standard goniometer will be used to measure patient range of motion for flexion, extension, side bending, and rotation. All measures will be completed in sitting and repeated two times in each direction. The standard error of measure for goniometry is 2.4 to 4.9 degrees

SECONDARY OUTCOMES:
The Numerical Pain Rating System (NPRS) | Baseline, 3 weeks, 6 weeks, 3 months
  Used to measure the patients' pain and headache intensity. The NPRS is an 11-point scale where 0 designates 'No pain' and 10 designates 'The worst pain imaginable'.
Optimal Screening for Prediction of Referral and Outcome-Yellow Flag (OSPRO-YF) | Baseline, 3 weeks, 6 weeks, 3 months
  The OSPRO-YF informs treatment decision-making and facilitates treatment monitoring for patients determined to be at high risk for poor outcomes by existing risk-assessment tools. The 10-item version has been found to have an accuracy of 81% in identifying yellow flags
The Neck Disability Index (NDI) | Baseline, 3 weeks, 6 weeks, 3 months
  A self-reported disability measure used in the study. A 5.5-point reduction in NDI score would deem the treatment clinically meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Borgehammar, DSc, Study Director — Midwestern University
Locations (2):
- United States (2):
  - Center for Orthopedic & Sports Physical Therapy, Tallahassee, Florida
  - OrthoPT Spine & Joint Specialists Clinic, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided
If data is shared it would be deidentified data reported in aggregate format only.

REFERENCES:
- [Result] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Result] Ritchie C, Sterling M. Recovery Pathways and Prognosis After Whiplash Injury. J Orthop Sports Phys Ther. 2016 Oct;46(10):851-861. doi: 10.2519/jospt.2016.6918. Epub 2016 Sep 3. PMID 27594661
- [Result] Ritchie C, Hendrikz J, Jull G, Elliott J, Sterling M. External validation of a clinical prediction rule to predict full recovery and ongoing moderate/severe disability following acute whiplash injury. J Orthop Sports Phys Ther. 2015 Apr;45(4):242-50. doi: 10.2519/jospt.2015.5642. PMID 25827122
- [Result] Garcia AN, Costa LDCM, de Souza FS, de Almeida MO, Araujo AC, Hancock M, Costa LOP. Reliability of the Mechanical Diagnosis and Therapy System in Patients With Spinal Pain: A Systematic Review. J Orthop Sports Phys Ther. 2018 Dec;48(12):923-933. doi: 10.2519/jospt.2018.7876. Epub 2018 Jun 22. PMID 29932871
- [Result] Jull GA, O'Leary SP, Falla DL. Clinical assessment of the deep cervical flexor muscles: the craniocervical flexion test. J Manipulative Physiol Ther. 2008 Sep;31(7):525-33. doi: 10.1016/j.jmpt.2008.08.003. PMID 18804003
- [Result] Domenech MA, Sizer PS, Dedrick GS, McGalliard MK, Brismee JM. The deep neck flexor endurance test: normative data scores in healthy adults. PM R. 2011 Feb;3(2):105-10. doi: 10.1016/j.pmrj.2010.10.023. PMID 21333948